CLINICAL TRIAL: NCT04421274
Title: Bone Marrow Mesenchymal Stem Cells Transfer in Patients With ST-segment Elevation Myocardial Infarction: Single-blind, Randomized Controlled Muticentre Trial
Brief Title: Bone Marrow Mesenchymal Stem Cells Transfer in Patients With ST-segment Elevation Myocardial Infarction
Acronym: Bmmsct
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Collaborators: Chinese PLA General Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ScPHFPC-100306
Record Dates: First submitted 2020-05-14; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Mesenchymal stem cells; Bone marrow; Stem cells transplantation
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BM-MSCs group (Experimental): Receive the best medication, percutaneous coronary intervention, and bone marrow mesenchymal stem cells transfer(Intracoronary artery )
  Interventions: Biological: Bone marrow mesenchymal stem cells transfer; Drug: Best medical treatment; Procedure: Percutaneous coronary intervention
- Control group (Sham Comparator): Receive the best medication, percutaneous coronary intervention
  Interventions: Drug: Best medical treatment; Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Biological: Bone marrow mesenchymal stem cells transfer — Inject the BM-MSCs into the infarct-related arterial hypertension through the central cavity of the guide wire balloon catheter under the complete blockage of the target blood vessel. Each time the balloon continues to fill for 2 minutes to block blood flow, then resume perfusion for 2 minutes. The above process is repeated 6 ~ 8 times
  Arms: BM-MSCs group
Drug: Best medical treatment — Refer to the latest medication guidelines and give the best medication to the patients
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention

SUMMARY:
To investigate the effect and safety of intracoronary autologous bone morrow mesenchymal stem cells (BM-MSCs) transplantation in patients with ST-segment elevation myocardial infarction（ STEMI） .

DETAILED DESCRIPTION:
To investigate the safety of intra-coronary injection of autologous bone marrow mesenchymal stem cells (BM-MSCs) in patients with ST-segment elevation myocardial infarction and its effect on cardiac function and viable myocardium. We plan to include approximately 40 patients with ST-segment elevation myocardial infarction as a research object, and conduct a randomized, single-blind, parallel-controlled multi-center clinical trial. The patients were randomly divided into a BM-MSCs group and a control group, and were given the best drug treatment and percutaneous coronary intervention (PCI). The primary study endpoint was the change in myocardial metabolic activity 6 months after autologous BM-MSCs transplantation and the change in left ventricular ejection fraction (LVEF) at 12 months; The incidence of adverse events. The above indexes were evaluated by cardiac color echocardiography and single photon emission computed tomography (SPECT).

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old;
* Diagnosed acute ST-elevation myocardial infarction (STEMI)
* STEMI onset <1 month
* Successful vascular remodeling, blood flow of infarct-related blood vessels recovered to TIMI level 3
* All patients included in the study signed an informed consent form and promised to complete all follow-up plans

Exclusion Criteria:

* Refractory persistent ventricular tachycardia
* High cardiac block and no pacemaker control
* Liver or renal dysfunction (ALT>80U/ L, Cr> 440mmol / L)
* Bleeding disorders, malignant tumors
* Autoimmune disease or any serious fatal disease
* Contraindications for coronary intervention
* Combined with other heart disease: congenital heart Disease (ventricular deficiency, atrial deficient, patent ductus arteriosus and other congenital alformations),primary valvular disease, active myocarditis, pulmonary heart disease,hyperthyroidism, mucous edema heart disease and so on
* Mental illness, no self-awareness, and no precise expression and cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2010-07-10 (Actual); Study Completion 2011-07-15 (Actual)

PRIMARY OUTCOMES:
changes in myocardial metabolic activity | Baseline + after 6 months
  changes in myocardial metabolic activity 6 months after transplantation of autologous BM-MSCs (SPET assay)
Changes in left ventricular ejection fraction (LVEF) | Baseline + after 12 months
  Changes in left ventricular ejection fraction (LVEF) at 12 months after transplantation of autologous BM-MSCs.

SECONDARY OUTCOMES:
incidence of cardiovascular events | in 12 months after transplantation of autologous BM-MSCs
  incidence of cardiovascular events
overall mortality | in 12 months after transplantation of autologous BM-MSCs
  overall mortality
adverse events at 12 months after transplantation of autologous BM-MSCs | in 12 months after transplantation of autologous BM-MSCs
  adverse events at 12 months after transplantation of autologous BM-MSCs

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Mianyang, Mianyang, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Unfortunately, the research data is not shared

REFERENCES:
- [Derived] Zhang R, Yu J, Zhang N, Li W, Wang J, Cai G, Chen Y, Yang Y, Liu Z. Bone marrow mesenchymal stem cells transfer in patients with ST-segment elevation myocardial infarction: single-blind, multicenter, randomized controlled trial. Stem Cell Res Ther. 2021 Jan 7;12(1):33. doi: 10.1186/s13287-020-02096-6. PMID 33413636